CLINICAL TRIAL: NCT02095444
Title: Phase1 Study of Recombinant Stem Cells That Repair Lung Injury in H7N9 Infected Patients
Brief Title: Using Human Menstrual Blood Cells to Treat Acute Lung Injury Caused by H7N9 Bird Flu Virus Infection
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: S-Evans Biosciences Co., Ltd. (Industry)
Collaborators: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEB-2014-2-20
Record Dates: First submitted 2014-03-16; First posted 2014-03-24 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Acute Lung Injury; Acute Respiratory Distress Syndrome (ARDS); Multiple Organ Failure
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome; Multiple Organ Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Menstrual blood stem cells (Experimental): 1x10*7 cells/kg, IV(in the vein) twice a week. Number of course for two weeks.
  Interventions: Drug: Menstrual blood stem cells

INTERVENTIONS:
Drug: Menstrual blood stem cells — 10*7 cells/kg, intravenous injection for 4 times during two weeks

SUMMARY:
The purpose of this study is to determine whether human menstrual blood-derived stem cells are effective in the treatment of infection of H7N9 virus caused acute lung injury.

DETAILED DESCRIPTION:
1. recruiting volunteers of H7N9 infection: age > 18; patients signed with the informed consent; APACHE II > 20 score
2. patients infused with menstrual blood progenitor cells infusion dose: 1~10×10*7 cells/kg infusion frequency: 2 times a week, 2 weeks for infusion
3. test items and standard spirits lifted; pulmonary function improved; lung image injury improved

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of H7N9 infection
* must be critical injured for lung tissues

Exclusion Criteria:

* cancer diseases
* pregnancy
* mental disorder
* allergic constitution
* severe inflammation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The degree of lung injury | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Xiang, Doctor, Principal Investigator — State Key Laboratory for Diagnosis and Treatment of Infectious Diseases, the First Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- State Key Laboratory for Diagnosis and Treatment of Infectious Diseases, the First Affiliated Hospital, Hangzhou, Zhejiang, China